CLINICAL TRIAL: NCT00341809
Title: Role of HLA and KIR in the Natural History of Psoriasis
Brief Title: Genetic Analysis of Psoriasis and Psoriatic Arthritis
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904255; 04-C-N255
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2012-09-04

CONDITIONS: Psoriasis
Keywords: Natural Killer Cells; Autoimmune Disease; Chronic Inflammation; Two-Locus Interaction; Allele/Haplotype Analysis
MeSH Terms: conditions — Psoriasis; Autoimmune Diseases

SUMMARY:
This study will examine the genetic basis of psoriasis and psoriatic arthritis. It is known that genes play an important role in determining who gets psoriasis or psoriatic arthritis. This study will look for specific gene variants (alleles) that run in families with these conditions, or are found more often in people with these conditions than in those without them.

Participants for this study were identified through the dermatology services of the University of Michigan Medical Center, the Ann Arbor Veterans Affairs Medical Center, the University of Kiel, and Henry Ford Hospital. Additional families were provided by the National Psoriasis Foundation Tissue Bank. They include people with psoriasis or psoriatic arthritis, or both, in addition to some family members of patients. Only families in which the age of the patient at disease onset was below 40 years are included. Patients were included if they had lesions covering more than 1 percent of their total body surface area or if at least two skin, scalp, nail, or joint lesions were diagnosed as psoriasis. Healthy volunteers are also enrolled as control subjects.

Participants undergo the following procedures, as follows:

Patients with psoriasis and people without psoriasis who have multiple family members with the disease

* Skin evaluation
* Photographs of lesions for documentation

Patients with psoriatic arthritis and people without psoriatic arthritis who have multiple family members with the disease

* Joint evaluation and possibly ultrasound
* Joint X-rays or review of existing X-rays

Patients with psoriasis only, with psoriatic arthritis, and healthy volunteers

* Blood draw of 30 milliliters. Some of the blood collected will be used to test for rheumatoid factor and C-reactive protein in patients with psoriatic arthritis.
* Periodic questionnaires to update health status information

DETAILED DESCRIPTION:
The aim of the study is to examine the role of HLA and killer immunoglobulin-like receptors (KIR) in the natural history of psoriasis vulgaris. Psoriasis is a chronic inflammatory disease of the skin with features of an autoimmune disease, and previous studies have revealed an association with certain HLA class I alleles, notably HLA-Cw*0602. Natural Killer (NK) cells are a unique group of lymphocytes involved in surveillance of killing of foreign or infected cells through a mechanism involving recognition of HLA class I molecules by an extremely diverse set of receptors on the NK cell surface. A major group of these receptors are the KIRs. Thus, a relationship between KIR/HLA genotype and psoriasis is biologically plausible, and indeed previous data from our laboratory have shown a strong association with the activating genes KIR2DS1 and KIR2DS2 and development of psoriatic arthritis, a well-recognized complication of psoriasis.

Dr. James Elder and colleagues at the University of Michigan have identified a cohort of more than 560 families through the dermatology services of the University of Michigan Medical Center, the University of Kiel, Henry Ford Hospital, and the National Psoriasis Foundation Tissue Bank. Individuals have been well characterized clinically, and information on race, ethnicity, age at onset, current age, and history of inflammatory bowel disease and/or other autoimmune disorders has been obtained. The large size of the cohort will provide substantial statistical power, which is of major importance in any KIR/HLA association study.

ELIGIBILITY:
* INCLUSION CRITERIA:

DNA and relevant clinical data from properly consented subjects will be provided to the LGD for genotyping and analysis. No available subjects will be excluded.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2653 (Actual)
Dates: Start 2004-07-30; Study Completion 2012-09-04

CONTACTS AND LOCATIONS:
Overall Officials: Michael Dean, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- [Background] Elder JT, Nair RP, Guo SW, Henseler T, Christophers E, Voorhees JJ. The genetics of psoriasis. Arch Dermatol. 1994 Feb;130(2):216-24. PMID 8304761
- [Background] Bhalerao J, Bowcock AM. The genetics of psoriasis: a complex disorder of the skin and immune system. Hum Mol Genet. 1998;7(10):1537-45. doi: 10.1093/hmg/7.10.1537. PMID 9735374
- [Background] Nair RP, Henseler T, Jenisch S, Stuart P, Bichakjian CK, Lenk W, Westphal E, Guo SW, Christophers E, Voorhees JJ, Elder JT. Evidence for two psoriasis susceptibility loci (HLA and 17q) and two novel candidate regions (16q and 20p) by genome-wide scan. Hum Mol Genet. 1997 Aug;6(8):1349-56. doi: 10.1093/hmg/6.8.1349. PMID 9259283